CLINICAL TRIAL: NCT06025045
Title: Dynamic Monitoring of ctDNA Predicts Recurrence of Advanced Ovarian Cancer After Primary Treatments
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jing Li (Other)
Collaborators: Nanjing Shihejiyin Technology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jing Li, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Other Study IDs: SunYatsen202309
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer Stage IV; Ovarian Cancer Stage III
Keywords: ctDNA; Ovarian cancer; PDS; IDS; adjuvant chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma sample； tumor tissue; WBC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who receive satisfactory PDS, currently the change in CA125 during chemotherapy can only be used to evaluate the effectiveness of chemotherapy. This study plans to use ctDNA dynamic monitoring to detect minimal residual lesions during treatment, to demonstrate the application value of ctDNA dynamic monitoring in predicting the recurrence of ovarian cancer after PDS/IDS surgery.

DETAILED DESCRIPTION:
This study plans to include ovarian cancer patients who have undergone PDS/IDS surgery. By analyzing the surgical tissue samples of ovarian cancer patients, we aim to identify risk factors related to the prognosis and recurrence of ovarian cancer. By monitoring the ctDNA status after PDS surgery, we analyze the role of ctDNA-MRD in predicting postoperative recurrence of ovarian cancer. By monitoring the MRD status at the end of the 3rd cycle of adjuvant chemotherapy and at the end of adjuvant treatment, we analyze the predictive role of serial cDNA-MRD for the efficacy of adjuvant treatment, providing a basis for determining the number of cycles of adjuvant treatment after PDS.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old.
2. Patients diagnosed with stage IIIC-IVA ovarian cancer through pathological examination.
3. The participant has read and fully understands the patient information, and has signed the informed consent form.
4. The patient is willing to undergo primary debulking surgery (PDS) or interval debulking surgery（IDS）. -

Exclusion Criteria:

1. Other tumors have been detected within the last 5 years.
2. Organ transplant recipients or those who previously had non-autologous (allogeneic) bone marrow or stem cell transplants.
3. Patients was deemed unsuitable to participate in this study by other researchers.
4. Patients who have previously received neoadjuvant chemotherapy or targeted therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced ovarian cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
2 years DFS rate | 2 years
  The recurrence rate of patients at two years after surgery

SECONDARY OUTCOMES:
DFS | 2 years
  Disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China